CLINICAL TRIAL: NCT03085901
Title: Comparison of Clinical Outcomes of Toric Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, tae-young chung, Professor, Samsung Medical Center, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-04-147
Record Dates: First submitted 2017-03-11; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precizon toric intraocular lens (Active Comparator): Cataract surgery and implantation of Precizon toric intraocular lens
  Interventions: Device: Precizon toric intraocular lens
- Tecnis toric intraocular lens (Active Comparator): Cataract surgery and implantation of Tecnis toric intraocular lens
  Interventions: Device: Tecnis toric intraocular lens

INTERVENTIONS:
Device: Precizon toric intraocular lens — Phacoemulsification and implantation of Precizon toric intraocular lens
  Arms: Precizon toric intraocular lens
Device: Tecnis toric intraocular lens — Phacoemulsification and implantation of Tecnis toric intraocular lens
  Arms: Tecnis toric intraocular lens

SUMMARY:
This study is to compare the clinical outcome of Precizon toric intraocular lens(IOL) to that of Tecnis toric IOL.

DETAILED DESCRIPTION:
In cataract surgery, after phacoemulsification, intraocular lens should be implanted for patient's better visual acuity. When patient has large amount of corneal astigmatism, toric intraocular lens are recommended to correct the preexisting astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cataract and regular corneal astigmatism(between 0.50 diopter and 2.50 diopter considering both anterior and posterior corneal surface)

Exclusion Criteria:

* Amblyopia, irregular astigmatism, corneal opacity, glaucoma, retinal disease, history of ocular inflammation, previous other intraocular surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Postoperative refractive astigmatism | postoperative 3 months
  Diopter

SECONDARY OUTCOMES:
Postoperative visual acuity | postoperative 3 months
  logMAR

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung NY, Lim DH, Hwang SS, Hyun J, Chung TY. Comparison of clinical outcomes of toric intraocular lens, Precizon vs Tecnis: a single center randomized controlled trial. BMC Ophthalmol. 2018 Nov 9;18(1):292. doi: 10.1186/s12886-018-0955-3. PMID 30413154